CLINICAL TRIAL: NCT05022043
Title: At Admission Serum Presepsin as Early Predictor for Disease Severity and Positive Blood Culture for Neonates With Early-onset Sepsis
Brief Title: Serum Presepsin as Early Predictor for Neonatal Early-onset Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed B.Hamza, lecturer of pediatrics and neonatology, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 34817/7/21
Record Dates: First submitted 2021-08-21; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Neonatal Sepsis
Keywords: Early-onset neonatal sepsis; Presepsin; Clinical scoring; Early predictors; Blood culture
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOS (Active Comparator)
  Interventions: Diagnostic Test: Serum Presepsin
- NO-EOS (No Intervention)

INTERVENTIONS:
Diagnostic Test: Serum Presepsin — Estimation of Serum Presepsin at time of admission
  Arms: EOS

SUMMARY:
124 neonates aged ≤7 days with suspected EOS were clinically evaluated using SNAP-II and gave blood samples for BC, total leucocytic count (TLC), lymphocytic and neutrophil count, and ELISA estimation of serum levels of PSP, procalcitonin (PCT), and tumor necrosis factor-α (TNF-α). Enrolled neonates were categorized as Confirmed EOS: neonates with evident clinical sepsis manifestations and positive BC, Suspected EOS: neonates with evident clinical sepsis manifestations but had negative BC and No EOS included neonates free of evident clinical sepsis manifestations, had negative BC and showed no deterioration till 72-hr after admission.

ELIGIBILITY:
Inclusion Criteria:

* included gestational age (GA) of 28-41 weeks and 5-min APGAR score of ≥7, and neonatal age of <7 days

Exclusion Criteria:

* including small for gestational age, presence of a chromosomal abnormality, multiple congenital anomalies, genetic syndromes, history of premature rupture of membranes, chorioamnionitis, neonatal asphyxia, and missed inclusion criterion.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
prediction of neonatal outcome | one week
  Ability of Serum Presepsin to disseminate neonates with confirmed EOS

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No